CLINICAL TRIAL: NCT02387866
Title: A Phase 1, Single Ascending Dose, Open-label Study to Evaluate the Pharmacokinetics and Safety of AG-221 in Healthy Male Japanese Subjects Relative to Healthy Male Caucasian Subjects
Brief Title: PK and Safety Study of AG-221 in Healthy Male Japanese Subjects and Healthy Male Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AG-221-CP-001
Expanded Access: NCT03723057 (No longer available)
Record Dates: First submitted 2015-03-05; First posted 2015-03-13 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Pharmacokinetic; Healthy Volunteers; Male; Japanese; Caucasian; AG-221
MeSH Terms: interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50 mg AG-221 tablet (Experimental): 50 mg AG-221 tablet given by mouth with 240 mL of non-carbonated, room temperature water, under fasted conditions
  Interventions: Drug: AG-221
- 100 mg AG-221 tablet (Experimental): 100 mg AG-221 tablet given by mouth with 240 mL of non-carbonated, room temperature water, under fasted conditions
  Interventions: Drug: AG-221
- 300 mg AG-221 tablet (Experimental): 300 mg AG-221 tablet given by mouth with 240 mL of non-carbonated, room temperature water, under fasted conditions
  Interventions: Drug: AG-221

INTERVENTIONS:
Drug: AG-221

SUMMARY:
This is a single ascending dose, open-label study that will evaluate the pharmacokinetics and safety of the AG-221 compound in normal, healthy volunteer male subjects (both Japanese and Caucasian).

DETAILED DESCRIPTION:
This is a phase 1, single ascending dose study to evaluate the PK and safety of AG-221 in healthy adult male Japanese subjects relative to healthy adult male Caucasian subjects. A total of 60 subjects will be enrolled; 30 will be Japanese subjects and 30 will be Caucasian subjects. There will be a total of 3 cohorts. Cohort A will receive a single dose of 100 mg AG-221. Cohort B will receive a single dose of 50 mg AG-221. Cohort C will receive a single dose of 300 mg AG-221. Within each cohort, 10 subjects will be Japanese and 10 subjects will be Caucasian.

Investigational product (IP) will be administered orally with approximately 240 mL of noncarbonated, room-temperature water. Subjects will enter the clinic prior to the evening meal on the day before dosing (Day -1) and will take a single oral dose of AG-221 at Hour 0 on the dosing day (Day 1), following a 10 hour overnight fast. After the dose is administered, subjects will be observed for 7 days to assess the acute safety profile before the next higher, protocol specified dose cohorts can enroll. The Sponsor and Investigator will review all available safety information prior to escalation to the next cohort to ensure that no safety issues exist.

Subjects will be confined to the study center from Day -1 to Day 3. Subjects will be discharged from the study center upon completion of the 48 hour PK blood draw. Subjects will return to the study center for additional PK blood draws on Days 5, 8, 11, 15, 22 and 29. In the event that a subject discontinues from the study, an early termination visit will be performed.

Blood samples will be collected at the following time (hours) for analysis of AG-221 and AGI-16903 (minor, active metabolite in humans) concentrations: Pre-dose, 1, 2, 3, 4, 6, 9, 12, 18, 24, 48, 96, 168, 240, 336, 504 and 672 hours.

In accordance with the guidance for clinical pharmacokinetic studies in Japan, this study design was selected to obtain PK data from Japanese in comparison to Caucasian healthy subjects. As the IP is an anticancer agent and, following the Japanese guidance for global studies, a single dose design was chosen.

AG-221 is a novel, first-in-class compound targeted specifically to inhibit the mutated IDH2 enzyme. AG-221 is currently being studied in a Phase 1 dose escalation study in subjects with advanced hematologic malignancies harboring an IDH2 mutation (AG221-C-001). The AG221-C-001 study is currently being conducted in the United States and France. This Japanese PK bridging study is intended to provide single dose PK and safety information in healthy Japanese subjects, relative to healthy Caucasian

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

Applicable to Japanese Subjects Only

1. Must have been born in Japan to both a Japanese mother and father and also have maternal and paternal Japanese grandparents.
2. Must understand and voluntarily sign an Informed Consent Form (ICF) written in English and Japanese prior to any study related procedures being performed and be able to adhere to restrictions and examination schedules.

Applicable to Caucasian Subjects Only

1. Must understand and voluntarily sign a written Informed Consent Form (ICF) prior to any study related procedures being performed and be able to adhere to restrictions and examination schedules.
2. Non-Japanese subjects must be Caucasian. Caucasian is defined as being of European or Latin American descent (ie, White).

Applicable to All Subjects

1. Healthy male subjects between 20 to 50 years of age (inclusive)
2. Must be able to communicate with the Investigator and understand and comply with the requirements of the study.
3. Must be in good health as determined by the Investigator according to past medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory tests.
4. Must have a body mass index (BMI) between 18 and 30 kg/m2 (inclusive).
5. Clinical laboratory tests must be within normal limits or considered by the Investigator to be not clinically significant.
6. Vital signs (systolic and diastolic blood pressure, pulse rate, and oral body temperature) will be assessed in the supine position after the subject has rested for at least 5 minutes. Subject must be afebrile (febrile is defined as ≥ 38 °C or 100.3° F) with vital signs within the following ranges:

   * Systolic blood pressure: 90 to 140 mm Hg
   * Diastolic blood pressure: 50 to 90 mm Hg
   * Pulse rate: 40 to 110 bpm
7. Must have a normal or clinically acceptable physical exam and 12-lead ECG. Subjects must have a QTcF value (Fridericia's Correction Factor) ≤ 450 msec. An ECG may be repeated up to 3 times to determine subject eligibility.
8. Subjects (with or without vasectomy) must agree to use barrier contraception (ie, latex condom or any synthetic material condom [eg, polyurethane] NOT made out of natural [animal] membrane) when engaging in sexual activity with women of childbearing potential (WCBP) while participating in the study. Subjects must refrain from sperm donations for the entire duration of the study.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Any serious medical condition, clinically significant laboratory abnormality, or psychiatric illness that would prevent the subject from signing the ICF and/or participating in the study.
  2. Recent history (ie, within 3 years prior to dosing) of any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological or other major disorders.
  3. Used any prescribed systemic or topical medication within 30 days of the first dose administration.
  4. Used any non-prescribed systemic or topical medication (including herbal medicines, eg, St. John's Wort) within 7 days of the first dose administration (with the exception of vitamin/mineral supplements).
  5. Subjects who have any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME) or subjects who plan to have any elective or medical procedures during the conduct of the trial.
  6. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
  7. Donated blood or plasma within 8 weeks preceding the first dose administration.
  8. History of multiple drug allergies (ie, 2 or more).
  9. Any clinically significant allergic disease.
  10. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years prior to dosing, or positive drug screening test due to illicit drugs.
  11. History of alcohol abuse within 2 years prior to dosing, or positive alcohol screen.
  12. Subjects who smoke more than 10 cigarettes or consume the equivalent in tobacco per day.
  13. Known to have hepatitis, or known to be a carrier of the HBsAg, or HCV Ab, or have a positive result to the test for HBsAg, HCV Ab, or HIV antibodies at Screening.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2015-05-21 (Actual); Study Completion 2015-07-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics -AUC 0-t | Up to 3 days
  Area under the plasma concentration-time curve from time zero to time t
Pharmacokinetics - AUC ∞ | Up to 3 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - Cmax | Up to 3 days
  Maximum observed plasma concentration
Pharmacokinetics - Tmax | Up to 3 days
  Time to maximum observed plasma concentration
Pharmacokinetics -T1/2 | Up to 3 days
  Estimate of the terminal elimination half-life in plasma
Pharmacokinetics -CL/F | Up to 3 days
  Apparent total plasma clearance when dosed orally
Pharmacokinetics -Vz/f | Up to 3 days
  Apparent volume of distribution during terminal phase

SECONDARY OUTCOMES:
Adverse Events (AEs) | Approximately 28 days
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene Corporation
Locations (1):
- Parexel International, Glendale, California, United States